CLINICAL TRIAL: NCT01125644
Title: Efficacy, Safety and Pharmacokinetics of SPK-843 in the Treatment of Pulmonary Mycosis. Open Label Phase III Clinical Study
Brief Title: Efficacy, Safety and Pharmacokinetics of SPK-843 in the Treatment of Pulmonary Mycosis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Proaparts srl (Industry)
Responsible Party: Tiberio Bruzzese, Proaparts srl
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPK-843-03/01
Record Dates: First submitted 2010-05-17; First posted 2010-05-18 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2011-06

CONDITIONS: Cryptococcosis or Aspergillosis Infections
Keywords: necrotic pulmonary infections
MeSH Terms: conditions — Cryptococcosis | interventions — SPA S 843

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single Arm (Experimental): Patients are males and females between 18 and 75 years of age with proven fungal etiology confirmed by mycological culture test and by hystopathological exam ("patients with definite diagnosis"), or patients with fungal infection of which is difficult to determine the etiological agent but with diagnosis of deep mycosis based on blood testing for fungal infection and/or clinical radiological examination, and/or endoscopic clinical examination, clinical symptomatology ("patients with clinical diagnosis").
  Interventions: Drug: SPK-843

INTERVENTIONS:
Drug: SPK-843 — SPK-843 is a semi-synthetic substance derived from Partricin A. 05 mg/Kg solution of SPK-843 in 10% intralipid will be administered i.v. in a hour for a treatment of 14 days
  Other Names: SPA-S-843

SUMMARY:
Recruitment of at least 10 adult patients (men and women) among individuals affected and admitted to the hospitals identified for the clinical study. All patients shall be between 18 and 75 years of age, with confirmed diagnosis of cryptococcosis or aspergillosis . During therapy (14 days) and examination (28 days), the patients will be subject to 7 doctor's visits (day 1,3,7,10,14,21, and 28).

DETAILED DESCRIPTION:
Objective: primary objective Evaluation of the overall global clinical response based on secondary end points from 1 to 6 at the end of the therapy (Study day 14) and at the final visit at the end of the study - follow-up- (Study day 28) in comparison to the initial clinical state.

The evaluation will be based on: improvement/normalization in relation to the semi-quantitative scales at 3, 4 and 5 items or at opinion expressed as positive for at least 3 of the first 6 secondary end points.

secondary objectives

1. Improvement on the basis of clinical symptoms;
2. Antifungal efficacy from the cultures;
3. Improvement on the basis of mycological blood testing;
4. Improvement on the basis of laboratory diagnosis (hemogasanalysis, ESR, CPR);
5. Improvement on the basis of radiological imaging (Rx, CAT HR,…);
6. Improvement on the basis of endoscopic examination;
7. Evaluate the plasma levels of SPK-843 after single dose and after multiple doses;
8. Evaluate the safety in the administration of SPK-843.

Methodology: Open label multi center study

ELIGIBILITY:
Inclusion Criteria:The following will be included in the study:

* Patients with proven fungal etiology confirmed by mycological culture test and by hystopathological exam ("patients with definite diagnosis"), or patients with fungal infection of which is difficult to determine the etiological agent but with diagnosis of deep mycosis based on blood testing for fungal infection and/or clinical radiological examination, and/or endoscopic clinical examination, clinical symptomatology ("patients with clinical diagnosis").
* Patients being treated with other anti-fungal drugs (i) showing a poor response to the treatment at least after 5 days of administration of the anti-fungal drug, (ii) that have had an adverse reaction to the drug prejudicing its use, determining the risk/benefit ratio unfavorable to the patient.
* Patients between 18 and 75 years of age.
* Patients able to understand the content of the Informed Consent and willing to participate in the study.
* Male and female patients.
* Patients initially admitted to the hospitals identified for this clinical study.
* Informed Consent.

Exclusion Criteria:

* Patients being treated with other anti-fungal drugs with improving clinical symptoms or with an unclear clinical course.
* Patients with intra-venous catheter and hospitalized with a diagnosis of fungemia but without clinical symptomatology twelve hours after the removal of the catheter.
* Patients with serious deep mycosis with low change of clinical efficacy (with a high probability of death event), or with serious concomitant illnesses or with complications, which may make difficult a safety evaluation of the treatment object of this study.
* Patients with a history of allergy to drugs like AMPH-B or with serious allergic reactions to drugs (shock after administration of drugs different from antifungals).
* Patients with serious hepatic, and/or renal, and/or cardiac failure or basic lung disease or with functionality of the organs with the following criteria:

  * AST (GOT) or ALT (GPT) higher five (5) times the highest normal value or 200 UI/L;
  * Blood creatinine higher than 2,0 mg/dl;
  * Proteinuira (qualitative test) 3+ or greater, or a total urinary excretion of proteins (quantitative test) of 3,5 g/day or higher;
  * Hyperkalemia or hypokalemia or with a basic level of sodium of 6,0 mEq/L or greater or less than 2,5 mEq/L;
  * Hyperlipidemia with a basic value of total cholesterol greater than 1,5 times the highest normal values or 300 mg/dl, triglycerides higher than twice the highest normal values or 300 mg/dl;
  * Patients that require the infusion of leucocytes;
  * Patients with arterial thrombosis or with serious coagulative dysfunctions;
  * Patients with diabetes mellitus associated with ketosis ;
  * Pregnant women or women who intend to become pregnant, women in purperium, or breast feeding;
  * Patients that participated in a clinical study (with any type of drugs, including anti-cancer drugs) or that have been recruited for observational clinical studies with pharmaceutical agents a month before the beginning of the treatment with SPK-843;
  * Patients who, according to the doctor, are not considered fit to be recruited in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2010-05; Primary Completion 2011-10 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the overall global clinical response | 28 days
  Evaluation of the overall global clinical response based on secondary end points from 1 to 6 at the end of the therapy (Study day 14) and at the final visit at the end of the study - follow-up- (Study day 28) in comparison to the initial clinical state.

SECONDARY OUTCOMES:
Evaluate the safety in the administration of SPK-843. | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Luigi Allegra, Ph.D., Study Director — Ospedale Maggiore di Milano IRCCS Policlinico; Francesco Blasi, MD, Principal Investigator — Ospedale Maggiore di Milano IRCCS Policlinico
Locations (1):
- Ospedale Maggiore di Milano IRCCS Policlinico Dipartimento Malattie Cardiovascolari e Respiratorie, Milan, Italy